# Evaluating the Occurrence of Engagement Patterns and Participation Trends Among Patients in Treatment Resistant Depression

This is an Informed Consent Form For Treatment Resistant
Depression Patients in <u>Power Clinical Trial's</u> Observational Study

Date: October 20, 2023

Introduction to This Informed Consent Form

If you are filling out this form, it indicates that you may be eligible to participate in a unique observational clinical study focusing on patients with treatment-resistant depression. This detailed guide covers the study's key aims, the research approach, and the impacts, which include both good and potentially negative effects. Before making a decision, it is critical to completely grasp the effects of your possible engagement, and getting counsel from your doctor can give vital insights. If any aspect of this text appears to be confusing or if you have any queries, please contact the researcher or the facilitator.

Understanding the Role of Clinical Trials in Treatment Resistant Depression

Treatment-resistant depression (TRD) refers to a condition where individuals with depression do not respond adequately to standard treatments, such as antidepressant medications or psychotherapy. It is a challenging and complex form of depression that requires a comprehensive evaluation and specialized care to address the symptoms effectively.

When individuals do not experience an improvement in their depressive symptoms after several trials of various antidepressant medications or therapies, they may be diagnosed with treatment-resistant depression. This condition can significantly impact the individual's quality of life, leading to persistent feelings of sadness, hopelessness, and a reduced ability to function in daily life.

Clinical trials focusing on treatment-resistant depression play a crucial role in evaluating the safety and efficacy of new treatments for this condition. These trials serve as indispensable tools in determining whether new medications outperform conventional therapies, providing strong evidence to endorse their broader adoption.

What distinguishes this particular study is its primary emphasis on the personal experiences of individuals dealing with treatment-resistant depression, actively participating in a clinical trial involving medical interventions. The key objective is to meticulously examine trial completion rates and voluntary withdrawals within this specific patient group.

## Importance of Observational Clinical Trials

Participating in this medical trial requires immersing oneself in an observational study, a critical component of this clinical research that is specifically designed to acquire insights through unobtrusive monitoring of patients as they continue to follow their treatment regimens.

Researchers will just follow your experience, thoroughly measuring the consequences of your condition and making no changes to your treatment. This trial design is critical for improving our understanding of the natural development of a certain medical condition and its impact on persons who are affected by it. Your voluntary participation in this observational study contributes to the progress of medical knowledge and the care delivered to persons with the same illness.

Setting This Study Apart from Other Treatment Resistant Depression Clinical Trials

Recognizing the distinctiveness of this research investigation is pivotal. It functions purely on an observational basis, signifying that your involvement will not include any specific therapies or interventions. To make an informed decision about potential

participation in a clinical trial, it is vital to comprehend the range of treatment resistant depression clinical research, including interventional studies where participants undergo diverse treatment regimens.

Making an educated choice regarding your future participation in a clinical trial needs an active approach comprising research and trial comparison. Clinicaltrials.gov and similar sites provide a wealth of information about <u>treatment resistant depression studies</u>. Furthermore, Power's specialist web platform offers a complete list of ongoing <u>treatment resistant depression clinical trials</u> that are currently recruiting volunteers. With rigorous study and a complete comprehension of the many clinical trial categories, you may confidently decide whether or not to participate.

## Protecting Your Anonymity in the Study

Maintaining the complete security of your data is critical during this study. To ensure your anonymity, you must refrain from entering any personal or identifiable information in your questionnaire replies. The committed research team is relentless in its dedication to improving privacy and security. However, it is critical to note that some legal scenarios may occur that require the disclosure of personal information.

## Actively Participating in Clinical Trial Surveys

We ask you to actively participate in this observational clinical study by contributing your views and experiences. Your involvement will entail completing surveys every two weeks, which will take around 20-30 minutes of your time. Furthermore, our staff is prepared to conduct quarterly check-in calls, guaranteeing continual support and involvement during the trial.

It is essential to highlight that your involvement in the survey phase of the trial is entirely voluntary. You have the option to select specific questions to respond to or complete the full questionnaire at your discretion. Furthermore, you maintain the right to withdraw from the trial at any time. Acknowledging the personal significance of enrolling in a clinical trial, we are committed to providing the necessary assistance, respecting your privacy, and guiding your decision-making process throughout the trial.

#### **Potential Benefits**

While participants in this observational clinical research may not see immediate advantages, their participation has the potential to have a long-term influence. The information gathered from participants will be useful in developing future ways for engaging persons suffering from treatment-resistant depression, possibly widening the landscape of medical research. Those who join this clinical trial have the potential to effect substantial improvements in the field of medical research, perhaps paving the way for future treatment-resistant depression patients.

## Potential Health Impacts and Risks

While clinical trials have resulted in important advances, it is critical to understand the possible health consequences that participants may suffer, especially in studies evaluating new drugs.

However, in observational clinical research, we use a special technique to minimize these effects by not administering experimental medications to subjects. Instead, our primary focus is on meticulous monitoring and assessment of outcomes, assuring the avoidance of any avoidable health hazards.

# **Enabling Diversity in Clinical Trials**

If you are interested in exploring the multifaceted nature of diversity in clinical trials, there are some online materials that you can read.

Whether you aim to understand the intricacies of the challenges and possibilities linked to clinical trial diversity or broaden your personal outlook, the following resources can be a valuable asset:

Rencsok, Emily M., Latifa A. Bazzi, Rana R. McKay, Franklin W. Huang, Adam Friedant, Jake Vinson, Samuel Peisch et al. "Diversity of enrollment in prostate cancer clinical trials: current status and future directions." *Cancer Epidemiology, Biomarkers & Prevention* 29, no. 7 (2020): 1374-1380.

<u>Bibbins-Domingo</u>, <u>Kirsten</u>, <u>Alex Helman</u>, <u>and Victor J. Dzau</u>. "The imperative for <u>diversity and inclusion in clinical trials and health research participation." *Jama* 327, no. 23 (2022): 2283-2284.</u>

## Confirmation of Understanding of Informed Consent

I confirm that I have spent enough time comprehending and internalizing the contents of the informed consent form. This comprehension was obtained by either independent review or with the assistance of research professionals who communicated its specifics to me. To my total pleasure, all of my issues and queries have been adequately answered.

I am fully aware that my participation in this study is purely voluntary, and I have the sole right to withdraw my permission without providing justifications or incurring any financial responsibilities. It has been made clear to me that a copy of this informed consent form will be supplied to me for my own records.

Following careful deliberation and a thorough assessment of all the information supplied to me, I hereby consent to participate in this study, indicating my informed and autonomous decision.

| Participant Name |
|-----------------------|
| Participant Signature |
| <br>Date |

Verification of Informed Consent Facilitator

I certify that I had a thorough discussion with the participant, thoroughly clarifying the complexities mentioned in this written paper. My goal was to ensure that the participant was completely aware of the primary research objectives, methodology used, potential risks and benefits, and other essential components of the treatment resistant depression clinical trial.

There was enough time for the participant to ask questions, voice concerns, and seek clarification. It is critical to emphasize that participation in this study is fully voluntary, and participants have the unlimited right to leave at any time, for any reason, without incurring any financial obligations.

Following the participant's permission, a properly kept copy of this written document, functioning as a repository for their personal information, was delivered.

| Printed Name of Assisting Researcher |
|--------------------------------------|
| Signature of Assisting Researcher |
| Date |